CLINICAL TRIAL: NCT05257005
Title: Natural History Study of Pyruvate Dehydrogenase Deficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: The Freya Foundation (Unknown); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 19GR12; 278183 (Other: Health Research Authority, United Kingdom); 283427 (Other: Health Research Authority, United Kingdom)
Record Dates: First submitted 2022-02-02; First posted 2022-02-25 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Pyruvate Dehydrogenase Complex Deficiency; Pyruvate Dehydrogenase E1 Alpha Deficiency; Pyruvate Dehydrogenase E1-Beta Deficiency; Pyruvate Dehydrogenase E2 Deficiency; Pyruvate Dehydrogenase Phosphatase Deficiency
Keywords: PDH deficiency; Natural History; Outcomes; Prognosis; Genotype-phenotype correlation; Quality of life; Outcome measures
MeSH Terms: conditions — Pyruvate Dehydrogenase Complex Deficiency Disease; Pyruvate Dehydrogenase E1 Alpha Deficiency; Pyruvate Dehydrogenase E1-Beta Deficiency; Pyruvate Dehydrogenase E2 Deficiency; Pyruvate dehydrogenase phosphatase deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient cohort: Non interventional study

SUMMARY:
Pyruvate dehydrogenase (PDH) deficiency is one of the most common mitochondrial disorders. Patients with this genetic condition have difficulty utilising carbohydrates to produce energy and develop a combination of problems including seizures, poor balance, developmental delay, disability and have a reduced life expectancy. As for most mitochondrial disorders there is a lack of effective treatments. It is essential to understand the mechanisms underlying the disease in order to identify new treatments, and to understand the natural history of disease in order to prepare for clinical trials. To date, a natural history study of PDH deficiency has not been undertaken in the UK.

The researchers aim to undertake the first natural history study of PDH deficiency in the UK, to describe the spectrum of symptoms, genetics, management and outcomes in both children and adult patients.

ELIGIBILITY:
Inclusion Criteria:

1. Compatible clinical history AND

2a Enzymatic confirmation demonstrating reduced PDH activity in patient cells or muscle tissue OR

2b Confirmed pathogenic mutation in a gene associated with primary PDH deficiency (PDHA1, PDHB, PDHX, PDP1, DLAT) OR

2c First degree relative with a confirmed pathogenic mutation causing primary PDH deficiency

Exclusion Criteria:

Patients with 'secondary PDH deficiency' that is patients who meet criteria 1 and 2a but who have received a genetic diagnosis which confirms pathogenic variants in a gene not associated with primary PDH deficiency.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and Adults with a diagnosis of (primary) Pyruvate Dehydrogenase Deficiency who are recruited from the community via tertiary healthcare services
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Newcastle Mitochondrial Disease Scale | Baseline
  Newcastle Paediatric and Adult Mitochondrial Disease Scale This is a validated scoring system for mitochondrial disease patients and measures severity of disease using multiple different clinical outcome measures and questionnaires. A higher score indicates greater disease severity.

OTHER OUTCOMES:
Mitochondrial Disease Phenotype | Baseline
  PDH deficiency Phenotype
Genetic Diagnosis | Baseline
  Molecular diagnosis
Medical History | Baseline
  Family history, past medical history
Disease timecourse | Baseline
  Onset, symptom debut, final outcome, follow-up.
Neuroimaging | Baseline
  MRI/MRS Head
Assessment of Neurophysiological outcome measures from source data | Baseline
  This is an observational retrospective from source data and may include the following neurophysiological measures: EMG, EEG, Nerve conduction Studies
Assessment of Cognitive and Developmental outcomes from source data | Baseline
  Retrospective assessments documented within source data for cognitive assessments that have occurred in the past in all patients.
Assessment of Cognitive and Developmental outcomes at baseline | Baseline
  For prospective component, cognitive assessments will be performed at baseline in adult patients only:
  Wechsler Test of Adult Reading (WTAR) test Symbol Search Speed of comprehension test
Assessment of biochemical outcome measures from source data | Baseline
  This is an observational retrospective from source data and may include the following biological outcome measures: EMG, EEG, Nerve conduction Studies: Blood and CSF lactate, pyruvate, amino acids, urine organic acids, PDH enzymology, OXPHOS studies, skeletal muscle histology
Management | Baseline
  Drug and non-drug treatments

CONTACTS AND LOCATIONS:
Overall Officials: Shamima Rahman, PhD, Study Director — Great Ormond Street Hospital NHS Foundation Trust
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phoenix C, Schaefer AM, Elson JL, Morava E, Bugiani M, Uziel G, Smeitink JA, Turnbull DM, McFarland R. A scale to monitor progression and treatment of mitochondrial disease in children. Neuromuscul Disord. 2006 Dec;16(12):814-20. doi: 10.1016/j.nmd.2006.08.006. Epub 2006 Nov 22. PMID 17123819
- [Background] Patel KP, O'Brien TW, Subramony SH, Shuster J, Stacpoole PW. The spectrum of pyruvate dehydrogenase complex deficiency: clinical, biochemical and genetic features in 371 patients. Mol Genet Metab. 2012 Jul;106(3):385-94. doi: 10.1016/j.ymgme.2012.03.017. PMID 22896851